CLINICAL TRIAL: NCT05825612
Title: Reverse Cascade Screening for Familial Hypercholesterolemia in Children and Adolescents in Northwest Greece
Brief Title: EPIRUS FH Reverse Cascade Screening
Status: Not yet recruiting | Type: Observational
Sponsor: Hellenic Atherosclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: EPIRUS-FH
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Familial Hypercholesterolemia
Keywords: children; adolescents; reverse cascade screening
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Next-generation sequencing for the genes encoding PCSK9, APOB, LDLR και LDLRAP1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heterozygous Familial Hypercholesterolemia: Children and adolescents with Heterozygous Familial Hypercholesterolemia.
- Homozygous Familial Hypercholesterolemia: Children and adolescents with Homozygous Familial Hypercholesterolemia.
- Unaffected (non-FH) individuals: Children and adolescents not carrying the investigated FH mutations

SUMMARY:
Familial hypercholesterolemia (FH) is the most common inherited metabolic disorder resulting in marked elevations in low-density lipoprotein cholesterol (LDL-C). If left untreated, lifelong exposure to elevated LDL-C leads to a substantially increased risk of premature cardiovascular disease as compared to the general population. Although FH adverse cardiovascular outcomes are potentially preventable through early identification of FH individuals and initiation of effective treatment, available evidence shows that FH is under-diagnosed and under-treated.

Childhood is the optimal period for FH screening, because due to minimal dietary and hormonal influences, LDL-C levels reflect predominantly the genetic component in children and are well suited to discriminate FH from other causes of elevated LDL-C. If FH remains untreated in this latent stage of the disease, individuals show a 10-fold increase of cardiovascular risk during early and middle adulthood. In this context, an effective approach for detecting FH would be a screening during childhood or in young adolescents in combination with reverse cascade screening of first-degree relatives of FH individuals.

EPIRUS-FH registry is a model program of reverse cascade screening for FH in children and adolescents in Northwest Greece that aims to increase public and physician awareness, strengthen the national registry of familial hypercholesterolemia (HELLAS-FH) and constitute the core for a national FH registry in children and adolescents in Greece.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C >160 mg/dL on two seperate measurements 3 months apart
* LDL-C >130 mg/dL + family history of premature coronary artery disease or hypercholesterolemia in one parent
* Children and adolescents on cholesterol-lowering medication

Exclusion Criteria:

* Refusal to sign the consent form and disagreement with the terms of participation.
* Any clinically significant disorder recognized at the time of the preliminary assessment, which in the judgment of the investigator would disqualify patient's participation in the study.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients genetically diagnosed with familial hypercholesterolemia (FH). Non-affected (non-FH) individuals as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Familial Hypercholesterolemia | Baseline
  Type of FH (Heterozygous FH, Homozygous FH). In the case of genetic diagnosis, what gene was affected (LDL receptor, Apolipoprotein B, PCSK9, LDLRAP1, other to be specified).
  Age at diagnosis of FH.

IPD SHARING:
Plan to Share IPD: No